CLINICAL TRIAL: NCT01200368
Title: A Phase 3, Randomized, Active-controlled, Double-blind Trial Evaluating The Safety, Tolerability, And Immunogenicity Of A 13-valent Pneumococcal Conjugate Vaccine Given With Dtap Compared To Open-label Dtap In Healthy Japanese Infants
Brief Title: Trial Evaluating a 13-valent Pneumococcal Conjugate Vaccine Given With Diphtheria, Tetanus, and Acellular Pertussis Vaccine (DTaP) in Healthy Japanese Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B1851056; B1851056; 6096A1-3024 (Other: Alias Study Number)
Record Dates: First submitted 2010-08-31; First posted 2010-09-13 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Healthy Subjects
Keywords: vaccine; pneumococcal conjugate
MeSH Terms: interventions — Diphtheria-Tetanus-acellular Pertussis Vaccines; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Experimental
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine (13vPnC); Biological: diphtheria, tetanus, and acellular pertussis vaccine (DTaP)
- 2 (Active Comparator): Active comparator
  Interventions: Biological: 7-valent pneumococcal conjugate vaccine (7vPnC); Biological: DTaP
- 3 (Active Comparator): Active comparator
  Interventions: Biological: DTaP

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine (13vPnC) — 0.5 mL per dose, 4 doses
  Arms: 1
Biological: diphtheria, tetanus, and acellular pertussis vaccine (DTaP) — 0.5 mL per dose, 4 doses
  Arms: 1
Biological: 7-valent pneumococcal conjugate vaccine (7vPnC) — 0.5 mL per dose, 4 doses
  Arms: 2
Biological: DTaP — 0.5 mL per dose, 4 doses
  Arms: 2
Biological: DTaP — 0.5 mL per dose, 4 doses
  Arms: 3

SUMMARY:
Subjects will be randomly assigned to 1 of 3 groups to receive the following vaccines: Group 1: 13-valent pneumococcal conjugate vaccine (13vPnC) and diphtheria, tetanus, and acellular pertussis vaccine (DTaP), Group 2: 7-valent pneumococcal conjugate vaccine (7vPnC) and DTaP, Group 3: DTaP alone. Group 3 subjects will also receive catch-up doses of Prevenar (commercial product of Prevenar in Japan) 13vPnC and 7vPnC will be blinded, and DTaP will be open-label. The main purpose of the study is to determine if the immune responses to 13vPnC are comparable to the immune responses to 7vPnC and if the immune responses to 13vPnC given with DTaP are comparable to those induced by DTaP given alone. In addition, the study aims to evaluate the side effects (safety profile) after vaccination of 13vPnC and 7vPnC when given with DTaP in healthy Japanese infants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 3 to 6 months of age at the enrollment.
* Available for the entire study period and whose parent/legal guardian can be reached by telephone.
* Healthy infant as determined by medical history, physical examination, and judgement of the investigator.

Exclusion Criteria:

* Previous vaccination with licensed or investigational pneumococcal, diphtheria, tetanus, or pertussis vaccines.
* A previous anaphylactic reaction to any vaccine or vaccine-related component.
* Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate any type of injection.
* History of culture-proven invasive disease caused by S pneumoniae (eg, meningitis, bacteremia, osteomyelitis, arthritis).
* Infant who is a direct descendant (child, grandchild) of the study site personnel.

Ages: 3 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 551 (Actual)
Dates: Start 2010-09-24 (Actual); Primary Completion 2011-11-30 (Actual); Study Completion 2011-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (32):
- Japan (32):
  - Sunrise Children's Clinic, Funabashi, Chiba
  - Sotobo Children's Clinic, Isumi, Chiba
  - Matsuyama Red Cross Hospital, Matsuyama, Ehime
  - Fukazawa Pediatric Clinic, Higashi-ku, Fukuoka-city, Fukuoka
  - National Hospital Organization Fukuyama Medical Center, Fukuyama, Hiroshima
  - National Hospital Organization Kure Medical Center, Kure, Hiroshima
  - Nakata pediatric clinic, Sapporo, Hokkaido
  - Watanabe Pediatric Allergy Clinic, Sapporo, Hokkaido
  - Furuta Children's Clinic, Sapporo, Hokkaido
  - Motomachi pediatric clinic, Sapporo, Hokkaido
  - Tenshi Hospital, Sapporo, Hokkaido
  - Yoshimoto Pediatrist Clinic, Kikuchi-gun, Kumamoto
  - Shiroko Clinic, Suzuka, Mie-ken
  - National Mie Hospital, Tsu, Mie-ken
  - National hospital Organization Mie Chuou Medical Center, Tsu, Mie-ken
  - Children's Enomoto Clinic, Kumagaya, Saitama
  - Shibuya Clinic, Kumagaya, Saitama
  - Sakiyama Children's Clinic, Fuchū, Tokyo
  - Okawa Children and Family Clinic, Ōta-ku, Tokyo
  - Seijo Sasamoto Pediatric And Allergy Clinic, Setagaya-ku, Tokyo
  - National Center for Child Health and Development, Setagaya-ku, Tokyo
  - Miyata Pediatric Clinic, Tachikawa-shi, Tokyo
  - Maehara Pediatric Clinic, Tama, Tokyo
  - Childrens Clinic of Kose, Kofu, Yamanashi
  - Medical Corporation Bunpoukai Amemiya Clinic, Koushu-shi, Yamanashi
  - Medical Corporation Seijinkai Takei Clinic, Tsuru-shi, Yamanashi
  - National Hospital Organization Fukuoka National Hospital, Fukuoka
  - Harada Clinic, Fukuoka
  - Hattori Pediatric Clinic, Kumamoto
  - Medical Corporation Seiaikai Seguchi Pediatric Clinic, Kumamoto
  - Medical Corporation Oukakai Sakuranbo Kodomo Clinic, Kumamoto
  - Momotaro Clinic, Okayama

REFERENCES:
- [Derived] Togashi T, Okada K, Yamaji M, Thompson A, Gurtman A, Cutler M, Aizawa M, Gruber WC, Scott DA. Immunogenicity and Safety of a 13-Valent Pneumococcal Conjugate Vaccine Given With DTaP Vaccine in Healthy Infants in Japan. Pediatr Infect Dis J. 2015 Oct;34(10):1096-104. doi: 10.1097/INF.0000000000000819. PMID 26121200

RESULTS

PARTICIPANT FLOW:
Groups:
- 13vPnC + DTaP: Participants at 3 to 6 months of age received a single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) subcutaneously followed by 2 single 0.5 mL doses of 13vPnC subcutaneously, 4 to 8 weeks after each previous dose (infant series) and a single 0.5 mL dose of 13vPnC subcutaneously at 12 to 15 months of age (toddler dose). A single 0.5 mL dose of diphtheria, tetanus, and acellular pertussis vaccine (DTaP) subcutaneously administered concomitantly with each 13vPnC dose.
- 7vPnC + DTaP: Participants at 3 to 6 months of age received a single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) subcutaneously followed by 2 single 0.5 mL doses of 7vPnC subcutaneously 4 to 8 weeks after each previous dose (infant series) and a single 0.5 mL dose of 7vPnC subcutaneously at 12 to 15 months of age (toddler dose). A single 0.5 mL dose of DTaP subcutaneously administered concomitantly with each 7vPnC dose.
- DTaP (Catch-up 7vPnC): Participants at 3 to 6 months of age received a single 0.5 mL DTaP dose subcutaneously followed by 2 single 0.5 mL DTaP doses subcutaneously, 4 to 8 weeks after each previous dose (infant series). Four to 6 weeks post-infant series, 2 single catch-up (CU) doses of 7vPnC (Prevenar) were administered subcutaneously, 4 to 6 weeks apart. A single 0.5 mL DTaP dose subcutaneously at 12 to 15 months of age (toddler dose) followed by a single CU dose of 7vPnC (Prevenar) subcutaneously 4 to 6 weeks post-toddler dose.
Period: Infant Series
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Started | 183 | 184 | 184
Vaccinated Dose 1 | 183 | 183 | 183
Vaccinated Dose 2 | 183 | 182 | 183
Vaccinated Dose 3 | 181 | 178 | 182
Completed | 180 | 178 | 178
Not Completed | 3 | 6 | 6
Not completed — Adverse Event | 2 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 2 | 2
Not completed — Did not meet entrance criteria | 0 | 1 | 0
Not completed — Randomized, not vaccinated | 0 | 1 | 1
Not completed — Other | 1 | 0 | 0
Period: After Infant Series
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Started | 180 | 178 | 178
Completed | 162 | 162 | 169
Not Completed | 18 | 16 | 9
Not completed — Adverse Event | 6 | 6 | 3
Not completed — Withdrawal by Subject | 10 | 8 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Other | 1 | 2 | 2
Period: Toddler Dose
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Started | 162 | 162 | 169
Completed | 162 | 159 | 168
Not Completed | 0 | 3 | 1
Not completed — Adverse Event | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP | DTaP (Catch-up 7vPnC) | Total
Number analyzed (Participants) | 183 | 184 | 184 | 551
Age, Continuous [Mean (Standard Deviation); unit: months] | 4.1 (0.97) | 4.1 (0.97) | 4.2 (0.96) | 4.1 (0.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 91 | 91 | 269
  Male | 96 | 93 | 93 | 282

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Level Greater Than or Equal to (>=) 0.35 Microgram Per Milliliter (mcg/mL) 1 Month After the Infant Series
Description: Percentage of participants achieving predefined antibody threshold >=0.35 mcg/mL along with the corresponding 95% confidence interval (CI) for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F and 19A) are presented. Exact 2-sided CI based on the observed proportion of participants. To demonstrate non-inferiority, for 6 additional serotypes in 7vPnC + DTaP group, the lowest response observed among the 7 common serotypes in the group was taken as reference.
Time Frame: 1 month after the infant series
Population: Evaluable infant immunogenicity population: eligible participants who received the vaccine to which they were randomized at all 3 doses, had blood drawn within the protocol-specified time frames, had at least 1 valid and determinate assay result after Dose 3 for the proposed analysis, and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 7vPnC + DTaP: Participants at 3 to 6 months of age received a single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) subcutaneously followed by 2 single 0.5 mL doses of 7vPnC subcutaneously, 4 to 8 weeks after each previous dose (infant series) and a single 0.5 mL dose of 7vPnC subcutaneously at 12 to 15 months of age (toddler dose). A single 0.5 mL dose of DTaP subcutaneously administered concomitantly with each 7vPnC dose.
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP
Number analyzed (Participants) | 177 | 176
percentage of participants
  4 | 100.0 [97.9 to 100.0] | 100.0 [97.9 to 100.0]
  6B | 97.7 [94.3 to 99.4] | 99.4 [96.9 to 100.0]
  9V | 100.0 [97.9 to 100.0] | 100.0 [97.9 to 100.0]
  14 | 100.0 [97.9 to 100.0] | 100.0 [97.9 to 100.0]
  18C | 100.0 [97.9 to 100.0] | 100.0 [97.9 to 100.0]
  19F | 98.9 [96.0 to 99.9] | 96.6 [92.7 to 98.7]
  23F | 97.7 [94.3 to 99.4] | 98.3 [95.1 to 99.6]
  1 | 100.0 [97.9 to 100.0] | 96.6 [92.7 to 98.7]
  3 | 99.4 [96.9 to 100.0] | 96.6 [92.7 to 98.7]
  5 | 99.4 [96.9 to 100.0] | 96.6 [92.7 to 98.7]
  6A | 98.3 [95.1 to 99.6] | 96.6 [92.7 to 98.7]
  7F | 100.0 [97.9 to 100.0] | 96.6 [92.7 to 98.7]
  19A | 100.0 [97.9 to 100.0] | 96.6 [92.7 to 98.7]
Statistical Analysis 1: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 4: Difference ([13vPnC + DTaP] - [7vPnC + DTaP]) in proportions, expressed as a percentage presented along with exact 2-sided 95 percent (%) confidence interval (CI); Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was greater than (>) -0.10; Percent difference = 0.0, 95% CI 2-sided [-2.2 to 2.1]
Statistical Analysis 2: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 6B: Difference ([13vPnC + DTaP] - [7vPnC + DTaP]) in proportions, expressed as a percentage presented along with exact 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = -1.7, 95% CI 2-sided [-5.2 to 1.1]
Statistical Analysis 3: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 9V: Difference ([13vPnC + DTaP] - [7vPnC + DTaP]) in proportions, expressed as a percentage presented along with exact 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 0.0, 95% CI 2-sided [-2.1 to 2.1]
Statistical Analysis 4: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 14: Difference ([13vPnC + DTaP] - [7vPnC + DTaP]) in proportions, expressed as a percentage presented along with exact 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 0.0, 95% CI 2-sided [-2.1 to 2.1]
Statistical Analysis 5: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 18C: Difference ([13vPnC + DTaP] - [7vPnC + DTaP]) in proportions, expressed as a percentage presented along with exact 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 0.0, 95% CI 2-sided [-2.1 to 2.1]
Statistical Analysis 6: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 19F: Difference ([13vPnC + DTaP] - [7vPnC + DTaP]) in proportions, expressed as a percentage presented along with exact 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 2.3, 95% CI 2-sided [-1.1 to 6.3]
Statistical Analysis 7: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 23F: Difference ([13vPnC + DTaP] - [7vPnC + DTaP]) in proportions, expressed as a percentage presented along with exact 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = -0.6, 95% CI 2-sided [-4.2 to 2.9]
Statistical Analysis 8: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 1: Difference ([13vPnC + DTaP] - [7vPnC + DTaP]) in proportions, expressed as a percentage presented along with exact 2-sided 95% CI. Difference in proportions was calculated using the serotype with the lowest proportion among the 7 common serotypes in the 7vPnC + DTaP group as reference; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 3.4, 95% CI 2-sided [0.9 to 7.3]
Statistical Analysis 9: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 3: Difference ([13vPnC + DTaP] - [7vPnC + DTaP]) in proportions, expressed as a percentage presented along with exact 2-sided 95% CI. Difference in proportions was calculated using the serotype with the lowest proportion among the 7 common serotypes in the 7vPnC + DTaP group as reference; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 2.9, 95% CI 2-sided [-0.2 to 6.7]
Statistical Analysis 10: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 5: Difference ([13vPnC + DTaP] - [7vPnC + DTaP]) in proportions, expressed as a percentage presented along with exact 2-sided 95% CI. Difference in proportions was calculated using the serotype with the lowest proportion among the 7 common serotypes in the 7vPnC + DTaP group as reference; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 2.9, 95% CI 2-sided [-0.2 to 6.7]
Statistical Analysis 11: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 6A: Difference ([13vPnC + DTaP] - [7vPnC + DTaP]) in proportions, expressed as a percentage presented along with exact 2-sided 95% CI. Difference in proportions was calculated using the serotype with the lowest proportion among the 7 common serotypes in the 7vPnC + DTaP group as reference; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 1.7, 95% CI 2-sided [-1.9 to 5.8]
Statistical Analysis 12: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 7F: Difference ([13vPnC + DTaP] - [7vPnC + DTaP]) in proportions, expressed as a percentage presented along with exact 2-sided 95% CI. Difference in proportions was calculated using the serotype with the lowest proportion among the 7 common serotypes in the 7vPnC + DTaP group as reference; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 3.4, 95% CI 2-sided [0.9 to 7.3]
Statistical Analysis 13: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 19A: Difference ([13vPnC + DTaP] - [7vPnC + DTaP]) in proportions, expressed as a percentage presented along with exact 2-sided 95% CI. Difference in proportions was calculated using the serotype with the lowest proportion among the 7 common serotypes in the 7vPnC + DTaP group as reference; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 3.4, 95% CI 2-sided [1.0 to 7.3]

2. Primary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody for 7 Common Serotypes 1 Month After the Infant Series
Description: Antibody geometric mean concentration (GMC) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) are presented. GMC (13vPnC) and corresponding 2-sided 95% confidence intervals (CI) were evaluated. Geometric means (GMs) were calculated using all participants with available data for the specified blood draw.
Time Frame: 1 month after the infant series
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP
Number analyzed (Participants) | 177 | 176
mcg/mL
  4 | 9.40 [8.48 to 10.41] | 11.54 [10.51 to 12.67]
  6B | 4.50 [3.90 to 5.21] | 5.71 [4.93 to 6.63]
  9V | 5.04 [4.52 to 5.62] | 6.80 [6.15 to 7.52]
  14 | 13.86 [12.16 to 15.80] | 16.79 [15.03 to 18.76]
  18C | 5.30 [4.75 to 5.91] | 7.26 [6.53 to 8.08]
  19F | 7.37 [6.43 to 8.46] | 8.38 [7.17 to 9.80]
  23F | 3.64 [3.16 to 4.19] | 4.53 [3.96 to 5.18]
Statistical Analysis 1: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 4: Ratio of IgG GMCs ([13vPnC + DTaP]/[7vPnC + DTaP]) was calculated along with 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for the IgG GMC ratio was >0.5; GMC ratio = 0.81, 95% CI 2-sided [0.71 to 0.94]
Statistical Analysis 2: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 6B: Ratio of IgG GMCs ([13vPnC + DTaP]/[7vPnC + DTaP]) was calculated along with 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 0.79, 95% CI 2-sided [0.64 to 0.97]
Statistical Analysis 3: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 9V: Ratio of IgG GMCs ([13vPnC + DTaP]/[7vPnC + DTaP]) was calculated along with 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 0.74, 95% CI 2-sided [0.64 to 0.86]
Statistical Analysis 4: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 14: Ratio of IgG GMCs ([13vPnC + DTaP]/[7vPnC + DTaP]) was calculated along with 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 0.83, 95% CI 2-sided [0.70 to 0.98]
Statistical Analysis 5: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 18C: Ratio of IgG GMCs ([13vPnC + DTaP]/[7vPnC + DTaP]) was calculated along with 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 0.73, 95% CI 2-sided [0.63 to 0.85]
Statistical Analysis 6: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 19F: Ratio of IgG GMCs ([13vPnC + DTaP]/[7vPnC + DTaP]) was calculated along with 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 0.88, 95% CI 2-sided [0.72 to 1.08]
Statistical Analysis 7: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 23F: Ratio of IgG GMCs ([13vPnC + DTaP]/[7vPnC + DTaP]) was calculated along with 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 0.80, 95% CI 2-sided [0.66 to 0.98]

3. Primary Outcome: Percentage of Participants Achieving Predefined Antibody Levels for Diphtheria Toxoid, Tetanus Toxoid, and Pertussis Antigens 1 Month After the Infant Series
Description: Predefined antibody levels were 0.1 International Units/mL (IU/mL) for diphtheria, 0.01 IU/mL for tetanus, 5 Enzyme-linked Immunosorbent Assay (ELISA) units/mL (EU/mL) for pertussis toxoid (PT), and 5 EU/mL for filamentous hemagglutinin (FHA).
Time Frame: 1 month after the infant series
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 177 | 176 | 175
percentage of participants
  Diphtheria | 99.4 [96.9 to 100.0] | 96.6 [92.7 to 98.7] | 100.0 [97.9 to 100.0]
  Tetanus | 100.0 [97.9 to 100.0] | 100.0 [97.9 to 100.0] | 100.0 [97.9 to 100.0]
  Pertussis toxoid (PT) | 99.4 [96.9 to 100.0] | 96.6 [92.7 to 98.7] | 100.0 [97.9 to 100.0]
  Filamentous hemagglutinin (FHA) | 99.4 [96.9 to 100.0] | 96.6 [92.7 to 98.7] | 100.0 [97.9 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC + DTaP vs DTaP (Catch-up 7vPnC); Difference in percentage of participants achieving predefined antibody levels for diphtheria toxoid and corresponding 2-sided 95% CI were calculated; Test type: Superiority or Other; Percent difference = -0.6, 95% CI 2-sided [-3.1 to 1.6]
Statistical Analysis 2: Comparison: 13vPnC + DTaP vs DTaP (Catch-up 7vPnC); Difference in percentage of participants achieving predefined antibody levels for tetanus toxoid and corresponding 2-sided 95% CI were calculated; Test type: Superiority or Other; Percent difference = 0.0, 95% CI 2-sided [-2.1 to 2.2]
Statistical Analysis 3: Comparison: 13vPnC + DTaP vs DTaP (Catch-up 7vPnC); Difference in percentage of participants achieving predefined antibody levels for pertussis toxoid and corresponding 2-sided 95% CI were calculated; Test type: Superiority or Other; Percent difference = -0.6, 95% CI 2-sided [-3.1 to 1.6]
Statistical Analysis 4: Comparison: 13vPnC + DTaP vs DTaP (Catch-up 7vPnC); Difference in percentage of participants achieving predefined antibody levels for filamentous hemagglutinin and corresponding 2-sided 95% CI were calculated; Test type: Superiority or Other; Percent difference = -0.6, 95% CI 2-sided [-3.1 to 1.6]

4. Secondary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody for 6 Additional Serotypes 1 Month After the Infant Series
Description: Antibody GMC for 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. GMC (13vPnC) and corresponding 2-sided 95% CIs were evaluated. GMs were calculated using all participants with available data for the specified blood draw. To demonstrate non-inferiority, for 6 additional serotypes in 7vPnC + DTaP group, the lowest GMC observed among the 7 common serotypes in the group was taken as reference.
Time Frame: 1 month after the infant series
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP
Number analyzed (Participants) | 177 | 176
mcg/mL
  1 | 8.14 [7.23 to 9.18] | 4.53 [3.96 to 5.18]
  3 | 4.90 [4.43 to 5.42] | 4.53 [3.96 to 5.18]
  5 | 4.64 [4.14 to 5.20] | 4.53 [3.96 to 5.18]
  6A | 4.71 [4.15 to 5.34] | 4.53 [3.96 to 5.18]
  7F | 8.26 [7.45 to 9.17] | 4.53 [3.96 to 5.18]
  19A | 8.56 [7.67 to 9.56] | 4.53 [3.96 to 5.18]
Statistical Analysis 1: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 1: Ratio of IgG GMCs ([13vPnC + DTaP]/[7vPnC + DTaP]) was calculated along with 2-sided 95% CI. GMC ratio was calculated using the serotype with the lowest GMC among the 7 common serotypes in the 7vPnC + DTaP group as reference; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 1.80, 95% CI 2-sided [1.50 to 2.15]
Statistical Analysis 2: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 3: Ratio of IgG GMCs ([13vPnC + DTaP]/[7vPnC + DTaP]) was calculated along with 2-sided 95% CI. GMC ratio was calculated using the serotype with the lowest GMC among the 7 common serotypes in the 7vPnC + DTaP group as reference; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 1.08, 95% CI 2-sided [0.92 to 1.28]
Statistical Analysis 3: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 5: Ratio of IgG GMCs ([13vPnC + DTaP]/[7vPnC + DTaP]) was calculated along with 2-sided 95% CI. GMC ratio was calculated using the serotype with the lowest GMC among the 7 common serotypes in the 7vPnC + DTaP group as reference; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 1.03, 95% CI 2-sided [0.86 to 1.22]
Statistical Analysis 4: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 6A: Ratio of IgG GMCs ([13vPnC + DTaP]/[7vPnC + DTaP]) was calculated along with 2-sided 95% CI. GMC ratio was calculated using the serotype with the lowest GMC among the 7 common serotypes in the 7vPnC + DTaP group as reference; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 1.04, 95% CI 2-sided [0.87 to 1.25]
Statistical Analysis 5: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 7F: Ratio of IgG GMCs ([13vPnC + DTaP]/[7vPnC + DTaP]) was calculated along with 2-sided 95% CI. GMC ratio was calculated using the serotype with the lowest GMC among the 7 common serotypes in the 7vPnC + DTaP group as reference; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 1.83, 95% CI 2-sided [1.54 to 2.16]
Statistical Analysis 6: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 19A: Ratio of IgG GMCs ([13vPnC + DTaP]/[7vPnC + DTaP]) was calculated along with 2-sided 95% CI. GMC ratio was calculated using the serotype with the lowest GMC among the 7 common serotypes in the 7vPnC + DTaP group as reference; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 1.89, 95% CI 2-sided [1.59 to 2.25]

5. Secondary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Level >=0.35 mcg/mL 1 Month After the Toddler Dose
Description: Percentage of participants achieving predefined antibody threshold >=0.35 mcg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. Exact 2-sided CI based on the observed proportion of participants. To demonstrate non-inferiority, for 6 additional serotypes in 7vPnC + DTaP group, the lowest response observed among the 7 common serotypes in the group was taken as reference.
Time Frame: 1 month after the toddler dose
Population: Evaluable toddler immunogenicity set:eligible participants who received vaccine to which they were randomized at all 4 doses,had blood drawn within specified time,had >=1 valid assay result after toddler dose for analysis,had no major protocol violation.N(number of participants analyzed)=participants with determinate IgG antibody level to serotype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP
Number analyzed (Participants) | 158 | 154
percentage of participants
  4 | 100.0 [97.7 to 100.0] | 100.0 [97.6 to 100.0]
  6B | 100.0 [97.7 to 100.0] | 100.0 [97.6 to 100.0]
  9V | 100.0 [97.7 to 100.0] | 100.0 [97.6 to 100.0]
  14 | 100.0 [97.7 to 100.0] | 100.0 [97.6 to 100.0]
  18C | 100.0 [97.7 to 100.0] | 100.0 [97.6 to 100.0]
  19F | 98.7 [95.5 to 99.8] | 99.4 [96.4 to 100.0]
  23F | 100.0 [97.7 to 100.0] | 100.0 [97.6 to 100.0]
  1 | 99.4 [96.5 to 100.0] | 99.4 [96.4 to 100.0]
  3 | 99.4 [96.5 to 100.0] | 99.4 [96.4 to 100.0]
  5 | 100.0 [97.7 to 100.0] | 99.4 [96.4 to 100.0]
  6A | 100.0 [97.7 to 100.0] | 99.4 [96.4 to 100.0]
  7F | 100.0 [97.7 to 100.0] | 99.4 [96.4 to 100.0]
  19A | 100.0 [97.7 to 100.0] | 99.4 [96.4 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 4: Difference ([13vPnC + DTaP] - [7vPnC + DTaP]) in proportions, expressed as a percentage presented along with exact 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 0.0, 95% CI 2-sided [-2.4 to 2.4]
Statistical Analysis 2: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 0.0, 95% CI 2-sided [-2.4 to 2.4]
Statistical Analysis 3: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; [analysis description as in outcome 1, analysis 3]; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 0.0, 95% CI 2-sided [-2.4 to 2.4]
Statistical Analysis 4: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; [analysis description as in outcome 1, analysis 4]; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 0.0, 95% CI 2-sided [-2.4 to 2.4]
Statistical Analysis 5: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; [analysis description as in outcome 1, analysis 5]; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 0.0, 95% CI 2-sided [-2.4 to 2.4]
Statistical Analysis 6: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; [analysis description as in outcome 1, analysis 6]; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = -0.6, 95% CI 2-sided [-3.9 to 2.4]
Statistical Analysis 7: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; [analysis description as in outcome 1, analysis 7]; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 0.0, 95% CI 2-sided [-2.4 to 2.4]
Statistical Analysis 8: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; [analysis description as in outcome 1, analysis 8]; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 0.0, 95% CI 2-sided [-2.9 to 3.0]
Statistical Analysis 9: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; [analysis description as in outcome 1, analysis 9]; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 0.0, 95% CI 2-sided [-2.9 to 3.0]
Statistical Analysis 10: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; [analysis description as in outcome 1, analysis 10]; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 0.6, 95% CI 2-sided [-1.7 to 3.6]
Statistical Analysis 11: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; [analysis description as in outcome 1, analysis 11]; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 0.6, 95% CI 2-sided [-1.7 to 3.6]
Statistical Analysis 12: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; [analysis description as in outcome 1, analysis 12]; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 0.6, 95% CI 2-sided [-1.7 to 3.6]
Statistical Analysis 13: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; [analysis description as in outcome 1, analysis 13]; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower confidence interval for the percent difference was >-0.10; Percent difference = 0.6, 95% CI 2-sided [-1.7 to 3.6]

6. Secondary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After the Toddler Dose
Description: Antibody GMC as measured by mcg/mL for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. GMC (13vPnC) and corresponding 2-sided 95% confidence intervals (CI) were evaluated. Geometric means (GMs) were calculated using all participants with available data for the specified blood draw. To demonstrate non-inferiority, for 6 additional serotypes in 7vPnC + DTaP group, the lowest GMC observed among the 7 common serotypes in the group was taken as reference.
Time Frame: 1 month after the toddler dose
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP
Number analyzed (Participants) | 158 | 154
mcg/mL
  4 | 15.34 [13.23 to 17.79] | 16.35 [14.19 to 18.83]
  6B | 17.05 [14.47 to 20.08] | 13.91 [11.93 to 16.21]
  9V | 7.00 [6.11 to 8.03] | 8.64 [7.54 to 9.89]
  14 | 19.70 [17.69 to 21.93] | 20.69 [18.25 to 23.47]
  18C | 8.10 [6.94 to 9.47] | 9.88 [8.64 to 11.30]
  19F | 16.73 [14.20 to 19.71] | 9.55 [8.11 to 11.26]
  23F | 8.64 [7.46 to 10.01] | 10.00 [8.61 to 11.62]
  1 | 13.96 [11.94 to 16.31] | 8.64 [7.54 to 9.89]
  3 | 2.48 [2.17 to 2.85] | 8.64 [7.54 to 9.89]
  5 | 11.10 [9.83 to 12.53] | 8.64 [7.54 to 9.89]
  6A | 15.17 [13.31 to 17.30] | 8.64 [7.54 to 9.89]
  7F | 10.90 [9.54 to 12.45] | 8.64 [7.54 to 9.89]
  19A | 16.02 [14.07 to 18.25] | 8.64 [7.54 to 9.89]
Statistical Analysis 1: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 4: Ratio of IgG GMCs ([13vPnC + DTaP]/[7vPnC + DTaP]) was calculated along with 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 0.94, 95% CI 2-sided [0.77 to 1.15]
Statistical Analysis 2: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 6B: Ratio of IgG GMCs ([13vPnC + DTaP]/[7vPnC + DTaP]) was calculated along with 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 1.23, 95% CI 2-sided [0.98 to 1.53]
Statistical Analysis 3: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 9V: Ratio of IgG GMCs ([13vPnC + DTaP]/[7vPnC + DTaP]) was calculated along with 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 0.81, 95% CI 2-sided [0.67 to 0.98]
Statistical Analysis 4: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 14: Ratio of IgG GMCs ([13vPnC + DTaP]/[7vPnC + DTaP]) was calculated along with 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 0.95, 95% CI 2-sided [0.81 to 1.12]
Statistical Analysis 5: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 18C: Ratio of IgG GMCs ([13vPnC + DTaP]/[7vPnC + DTaP]) was calculated along with 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 0.82, 95% CI 2-sided [0.67 to 1.01]
Statistical Analysis 6: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 19F: Ratio of IgG GMCs ([13vPnC + DTaP]/[7vPnC + DTaP]) was calculated along with 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 1.75, 95% CI 2-sided [1.39 to 2.21]
Statistical Analysis 7: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; Serotype 23F: Ratio of IgG GMCs ([13vPnC + DTaP]/[7vPnC + DTaP]) was calculated along with 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 0.86, 95% CI 2-sided [0.70 to 1.07]
Statistical Analysis 8: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 1.62, 95% CI 2-sided [1.31 to 1.99]
Statistical Analysis 9: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; [analysis description as in outcome 4, analysis 2]; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 0.29, 95% CI 2-sided [0.24 to 0.35]
Statistical Analysis 10: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; [analysis description as in outcome 4, analysis 3]; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 1.28, 95% CI 2-sided [1.07 to 1.54]
Statistical Analysis 11: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; [analysis description as in outcome 4, analysis 4]; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 1.76, 95% CI 2-sided [1.46 to 2.12]
Statistical Analysis 12: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; [analysis description as in outcome 4, analysis 5]; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 1.26, 95% CI 2-sided [1.04 to 1.52]
Statistical Analysis 13: Comparison: 13vPnC + DTaP vs 7vPnC + DTaP; [analysis description as in outcome 4, analysis 6]; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower limit of the 2-sided, 95% CI for IgG GMC ratio was >0.5; GMC ratio = 1.85, 95% CI 2-sided [1.54 to 2.24]

7. Secondary Outcome: Percentage of Participants Achieving Predefined Antibody Levels for Diphtheria Toxoid, Tetanus Toxoid, and Pertussis Antigens 1 Month After the Toddler Dose
Description: Predefined antibody level was 0.1 IU/mL for diphtheria, 0.01 IU/mL for tetanus, 5 EU/mL for PT, and 5 EU/mL for FHA.
Time Frame: 1 month after the toddler dose
Population: Evaluable toddler immunogenicity population. N (number of participants analyzed) = number of participants with determinate DTaP antibody level to serotype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 157 | 154 | 163
percentage of participants
  Diphtheria | 100.0 [97.7 to 100.0] | 100.0 [97.6 to 100.0] | 100.0 [97.8 to 100.0]
  Tetanus | 100.0 [97.7 to 100.0] | 100.0 [97.6 to 100.0] | 100.0 [97.8 to 100.0]
  Pertussis toxoid (PT) | 100.0 [97.7 to 100.0] | 100.0 [97.6 to 100.0] | 100.0 [97.8 to 100.0]
  Filamentous hemagglutinin (FHA) | 100.0 [97.7 to 100.0] | 100.0 [97.6 to 100.0] | 100.0 [97.8 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC + DTaP vs DTaP (Catch-up 7vPnC); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Percent difference = 0.0, 95% CI 2-sided [-2.4 to 2.3]
Statistical Analysis 2: Comparison: 13vPnC + DTaP vs DTaP (Catch-up 7vPnC); [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; Percent difference = 0.0, 95% CI 2-sided [-2.4 to 2.3]
Statistical Analysis 3: Comparison: 13vPnC + DTaP vs DTaP (Catch-up 7vPnC); [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; Percent difference = 0.0, 95% CI 2-sided [-2.4 to 2.3]
Statistical Analysis 4: Comparison: 13vPnC + DTaP vs DTaP (Catch-up 7vPnC); [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; Percent difference = 0.0, 95% CI 2-sided [-2.4 to 2.3]

8. Secondary Outcome: Geometric Mean Concentration (GMC) for Antigen-specific Diphtheria and Tetanus Antibodies 1 Month After the Infant Series
Description: GMC was measured in IU/mL and corresponding 2-sided 95% CI were evaluated for diphtheria and tetanus antibodies.
Time Frame: 1 month after the infant series
Population: Evaluable infant immunogenicity population: eligible participants who received the vaccine to which they were randomized at all 3 doses, had blood drawn within the protocol-specified time frames, had at least 1 valid and determinate assay result for the proposed analysis, and had no major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 177 | 176 | 175
IU/mL
  Diphtheria | 1.03 [0.94 to 1.12] | 1.10 [0.97 to 1.25] | 0.93 [0.86 to 1.02]
  Tetanus | 1.50 [1.31 to 1.70] | 1.37 [1.17 to 1.60] | 1.66 [1.50 to 1.83]
Statistical Analysis 1: Comparison: 13vPnC + DTaP vs DTaP (Catch-up 7vPnC); GMC ratio for diphtheria toxoid and corresponding 2-sided 95% CI were calculated; Test type: Superiority or Other; GMC ratio = 1.10, 95% CI 2-sided [0.97 to 1.24]
Statistical Analysis 2: Comparison: 13vPnC + DTaP vs DTaP (Catch-up 7vPnC); GMC ratio for tetanus toxoid and corresponding 2-sided 95% CI were calculated; Test type: Superiority or Other; GMC ratio = 0.90, 95% CI 2-sided [0.77 to 1.06]

9. Secondary Outcome: Geometric Mean Concentration (GMC) for Antigen-specific Acellular Pertussis Antibodies 1 Month After the Infant Series
Description: GMC was measured in EU/mL and corresponding 2-sided 95% CI were evaluated for PT and FHA antibodies.
Time Frame: 1 month after the infant series
Population: Evaluable infant immunogenicity population: eligible participants who received the vaccine to which they were randomized at all expected doses, had blood drawn within the protocol-specified time frames, had at least 1 valid and determinate assay result for the proposed analysis, and had no major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 177 | 176 | 175
EU/mL
  Pertussis toxoid (PT) | 66.12 [60.45 to 72.32] | 57.26 [49.23 to 66.60] | 67.64 [62.87 to 72.78]
  Filamentous hemagglutinin (FHA) | 62.30 [56.59 to 68.59] | 53.86 [47.27 to 61.37] | 67.48 [61.64 to 73.86]
Statistical Analysis 1: Comparison: 13vPnC + DTaP vs DTaP (Catch-up 7vPnC); GMC ratio for pertussis toxoid and corresponding 2-sided 95% CI were calculated; Test type: Superiority or Other; GMC ratio = 0.98, 95% CI 2-sided [0.87 to 1.10]
Statistical Analysis 2: Comparison: 13vPnC + DTaP vs DTaP (Catch-up 7vPnC); GMC ratio for filamentous hemagglutinin and corresponding 2-sided 95% CI were calculated; Test type: Superiority or Other; GMC ratio = 0.92, 95% CI 2-sided [0.81 to 1.05]

10. Secondary Outcome: Geometric Mean Concentration (GMC) for Antigen-specific Diphtheria and Tetanus Antibody 1 Month After the Toddler Dose
Description: GMC was measured in IU/mL and corresponding 2-sided 95% CI were evaluated for diphtheria and tetanus antibodies.
Time Frame: 1 month after the toddler dose
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 157 | 154 | 163
IU/mL
  Diphtheria | 2.65 [2.43 to 2.90] | 3.18 [2.94 to 3.45] | 2.63 [2.39 to 2.91]
  Tetanus | 2.90 [2.56 to 3.28] | 2.60 [2.29 to 2.95] | 2.89 [2.58 to 3.25]
Statistical Analysis 1: Comparison: 13vPnC + DTaP vs DTaP (Catch-up 7vPnC); GMC ratio for diphtheria toxoid and corresponding 2-sided 95% CI were calculated; Test type: Superiority or Other; GMC ratio = 1.01, 95% CI 2-sided [0.88 to 1.15]
Statistical Analysis 2: Comparison: 13vPnC + DTaP vs DTaP (Catch-up 7vPnC); GMC ratio for tetanus toxoid and corresponding 2-sided 95% CI were calculated; Test type: Superiority or Other; GMC ratio = 1.00, 95% CI 2-sided [0.85 to 1.19]

11. Secondary Outcome: Geometric Mean Concentration (GMC) for Antigen-specific Acellular Pertussis Antibody 1 Month After the Toddler Dose
Description: GMC was measured in EU/mL and corresponding 2-sided 95% CI were evaluated for PT and FHA antibodies.
Time Frame: 1 month after the toddler dose
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 157 | 154 | 163
EU/mL
  Pertussis toxoid (PT) | 144.46 [130.68 to 159.68] | 135.65 [124.16 to 148.21] | 150.21 [136.20 to 165.65]
  Filamentous hemagglutinin (FHA) | 143.68 [130.94 to 157.66] | 141.19 [129.20 to 154.30] | 180.31 [163.12 to 199.32]
Statistical Analysis 1: Comparison: 13vPnC + DTaP vs DTaP (Catch-up 7vPnC); GMC ratio for pertussis toxoid and corresponding 2-sided 95% CI were calculated; Test type: Superiority or Other; GMC ratio = 0.96, 95% CI 2-sided [0.84 to 1.11]
Statistical Analysis 2: Comparison: 13vPnC + DTaP vs DTaP (Catch-up 7vPnC); GMC ratio for filamentous hemagglutinin and corresponding 2-sided 95% CI were calculated; Test type: Superiority or Other; GMC ratio = 0.80, 95% CI 2-sided [0.70 to 0.91]

12. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions: Infant Series Dose 1 (3 to 6 Months of Age)
Description: Local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Redness and swelling were scaled as Any (redness or swelling present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (2.5 to 7.0 cm); Severe (> 7.0 cm). Participants may be represented in more than 1 category.
Time Frame: Within 7 days after Dose 1 of the infant series
Population: Safety population included all participants who received at least 1 dose of study vaccine. 'N' (number of participants analyzed)=participants reporting yes for at least 1 day or no for all days for any local reaction. 'n'=participants reporting yes for at least 1 day or no for all days for the specified local reaction for each group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 175 | 174 | 165
percentage of participants
  Redness- Any (n=171, 172, 165) | 58.5 | 55.8 | 10.3
  Redness- Mild (n=170, 172, 165) | 48.2 | 51.2 | 10.3
  Redness- Moderate (n=164, 166, 162) | 18.9 | 18.1 | 0.0
  Redness- Severe (n=161, 162, 162) | 0.0 | 0.6 | 0.0
  Swelling- Any (n=168, 168, 164) | 41.1 | 35.7 | 4.9
  Swelling- Mild (n= 168, 168, 164) | 38.1 | 31.5 | 4.9
  Swelling- Moderate (n=162, 165, 162) | 12.3 | 12.7 | 0.0
  Swelling- severe (n=161, 162, 162) | 0.0 | 0.6 | 0.0
  Tenderness- Any (n=163, 164, 162) | 13.5 | 6.1 | 1.2
  Tenderness- Significant (n=161, 162, 162) | 0.0 | 0.0 | 0.0
  Any local reaction (n=175, 174, 165) | 68.0 | 60.9 | 12.1

13. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions: Infant Series Dose 2 (4 to 8 Months of Age)
Description: as for outcome 12
Time Frame: Within 7 days after Dose 2 of the infant series
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 167 | 173 | 164
percentage of participants
  Redness- Any (n= 166, 168, 161) | 62.7 | 61.9 | 36.6
  Redness- Mild (n= 166, 167, 161) | 56.0 | 56.9 | 34.8
  Redness- Moderate (n= 157, 159, 156) | 26.1 | 27.0 | 8.3
  Redness- Severe (n= 157, 154, 154) | 0.0 | 0.0 | 0.0
  Swelling- Any (n= 160, 171, 162) | 48.1 | 50.9 | 24.1
  Swelling- Mild (n= 160, 170, 162) | 44.4 | 48.2 | 22.8
  Swelling- Moderate (n= 157, 157, 155) | 19.7 | 17.8 | 5.8
  Swelling- severe (n= 157, 154, 154) | 0.0 | 0.0 | 0.0
  Tenderness- Any (n= 159, 154, 155) | 14.5 | 4.5 | 1.9
  Tenderness- Significant (n= 157, 154, 154) | 0.6 | 0.0 | 0.0
  Any local reaction (n=167, 173, 164) | 71.3 | 67.1 | 40.2

14. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions: Infant Series Dose 3 (5 to 10 Months of Age)
Description: as for outcome 12
Time Frame: Within 7 days after Dose 3 of the infant series
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 171 | 163 | 160
percentage of participants
  Redness- Any (n= 168, 162, 156) | 53.6 | 51.2 | 23.1
  Redness- Mild (n= 167, 160, 156) | 47.3 | 43.1 | 21.8
  Redness- Moderate (n= 152, 154, 153) | 17.1 | 22.1 | 2.0
  Redness- Severe (n= 149, 152, 152) | 0.0 | 0.0 | 0.0
  Swelling- Any (n= 164, 157, 159) | 43.9 | 37.6 | 21.4
  Swelling- Mild (n= 164, 156, 159) | 42.1 | 34.0 | 20.1
  Swelling- Moderate (n= 150, 154, 153) | 10.7 | 14.9 | 2.6
  Swelling- severe (n= 149, 152, 152) | 0.0 | 0.0 | 0.0
  Tenderness- Any (n= 153, 155, 153) | 7.8 | 7.1 | 2.6
  Tenderness- Significant (n= 149, 152, 152) | 0.0 | 0.0 | 0.7
  Any local reaction (n=171, 163, 160) | 62.0 | 55.8 | 28.8

15. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions: Toddler Dose (12 to 15 Months of Age)
Description: as for outcome 12
Time Frame: Within 7 days after the toddler dose
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 153 | 152 | 151
percentage of participants
  Redness- Any (n= 148, 152, 149) | 62.2 | 57.2 | 34.9
  Redness- Mild (n= 148, 151, 148) | 50.0 | 47.7 | 28.4
  Redness- Moderate (n= 141, 139, 145) | 27.7 | 27.3 | 13.1
  Redness- Severe (n= 140, 136, 141) | 0.0 | 0.0 | 0.0
  Swelling- Any (n= 149, 144, 148) | 49.0 | 45.8 | 26.4
  Swelling- Mild (n= 147, 143, 146) | 42.9 | 42.0 | 22.6
  Swelling- Moderate (n= 143, 138, 146) | 16.8 | 18.8 | 13.0
  Swelling- severe (n= 140, 136, 141) | 0.0 | 0.0 | 0.0
  Tenderness- Any (n= 142, 140 ,142) | 14.1 | 10.0 | 5.6
  Tenderness- Significant (n= 140, 136, 141) | 0.7 | 0.0 | 0.0
  Any local reaction (n=153, 152, 151) | 68.6 | 61.8 | 37.1

16. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events: Infant Series Dose 1 (3 to 6 Months of Age)
Description: Systemic events (any fever >= 37.5 degrees Celsius [C], decreased appetite, irritability, increased sleep, decreased sleep, and hives [urticaria]) were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: Within 7 days after Dose 1 of infant series
Population: Safety population included all participants who received at least 1 dose of study vaccine. 'N'(number of participants analyzed)=participants reporting yes for at least 1 day or no for all days for any systemic reaction. 'n'=participants reporting yes for at least 1 day or no for all days for specified systemic reaction for each group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 177 | 174 | 172
percentage of participants
  Fever >=37.5,=<39 degrees C (n=168, 168, 165) | 36.3 | 33.9 | 21.8
  Fever >39,=<40 degrees C (n=161, 163, 162) | 0.6 | 1.2 | 0.6
  Fever >40 degrees C (n=161, 162, 162) | 0.0 | 0.0 | 0.0
  Decreased appetite (n=163, 163, 165) | 12.9 | 9.2 | 7.3
  Irritability (n=165, 164, 164) | 18.8 | 16.5 | 12.2
  Increased sleep (n=170, 165, 165) | 28.8 | 26.7 | 21.8
  Decreased sleep (n=164, 169, 167) | 18.3 | 21.3 | 13.8
  Hives- urticaria (n=161, 162, 162) | 3.1 | 1.2 | 0.0
  Use of antipyretic medication (n= 161, 162, 162) | 3.7 | 2.5 | 0.6
  Any systemic event (n=177, 174, 172) | 61.0 | 59.8 | 43.0

17. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events: Infant Series Dose 2 (4 to 8 Months of Age)
Description: Systemic events (any fever >= 37.5 degrees C, decreased appetite, irritability, increased sleep, decreased sleep, and hives [urticaria]) were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: Within 7 days after Dose 2 of infant series
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 170 | 169 | 166
percentage of participants
  Fever >=37.5, =<39 degrees C (n=166, 161, 155) | 36.7 | 36.6 | 21.9
  Fever >39, =<40 degrees C (n=158, 155, 154) | 1.9 | 3.9 | 0.6
  Fever >40 degrees C (n=157, 154, 154) | 0.0 | 0.0 | 0.0
  Decreased appetite (n=158, 159, 155) | 11.4 | 14.5 | 7.1
  Irritability (n=162, 155, 156) | 17.9 | 18.7 | 10.9
  Increased sleep (n=163, 158, 163) | 22.7 | 22.2 | 22.7
  Decreased sleep (n=161, 157, 157) | 18.6 | 12.1 | 12.1
  Hives- urticaria (n=157, 154, 154) | 2.5 | 1.3 | 1.9
  Use of antipyretic medication (n=160, 155, 154) | 3.1 | 4.5 | 1.3
  Any systemic event (n=170, 169, 166) | 61.2 | 57.4 | 44.6

18. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events: Infant Series Dose 3 (5 to 10 Months of Age)
Description: as for outcome 17
Time Frame: Within 7 days after Dose 3 of infant series
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 168 | 164 | 159
percentage of participants
  Fever >=37.5, =<39 degrees C (n=162, 161, 157) | 34.6 | 30.4 | 24.2
  Fever >39, =<40 degrees C (n=150, 152, 153) | 3.3 | 2.0 | 3.3
  Fever >40 degrees C (n=149, 152, 152) | 0.0 | 0.7 | 0.0
  Decreased appetite (n=152, 155, 154) | 9.9 | 9.7 | 5.8
  Irritability (n=154, 156, 154) | 17.5 | 14.7 | 11.7
  Increased sleep (n=151, 157, 154) | 20.5 | 20.4 | 14.9
  Decreased sleep (n= 154, 156, 153) | 18.2 | 12.8 | 9.8
  Hives- urticaria (n= 149, 152, 152) | 1.3 | 0.0 | 1.3
  Use of antipyretic medication (n=150, 153, 154) | 2.0 | 3.3 | 4.5
  Any systemic event (n=168, 164, 159) | 57.7 | 50.0 | 40.9

19. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events: Toddler Dose (12 to 15 Months of Age)
Description: as for outcome 17
Time Frame: Within 7 days after the toddler dose
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC + DTaP | 7vPnC + DTaP | DTaP (Catch-up 7vPnC)
Number analyzed (Participants) | 148 | 152 | 149
percentage of participants
  Fever >=37.5, =<39 degrees C (n=145, 146, 146) | 49.0 | 49.3 | 31.5
  Fever >39, =<40 degrees C (n=141, 136, 141) | 4.3 | 8.8 | 3.5
  Fever >40 degrees C (n=139, 137, 141) | 1.4 | 2.2 | 0.0
  Decreased appetite (n=143, 141, 143) | 19.6 | 19.9 | 9.8
  Irritability (n=143, 141, 144) | 18.2 | 21.3 | 16.7
  Increased sleep (n=145, 142, 143) | 18.6 | 17.6 | 16.1
  Decreased sleep (n=142, 137, 141) | 12.7 | 9.5 | 11.3
  Hives- urticaria (n=140, 136, 141) | 3.6 | 2.2 | 2.1
  Use of antipyretic medication (n=141, 138, 142) | 7.1 | 9.4 | 4.2
  Any systemic event (n=148, 152, 149) | 62.8 | 63.8 | 50.3

ADVERSE EVENTS:
Time Frame: AEs/SAEs: recorded from signing of informed consent form to completion of study. Participants recorded pre-specified AEs in electronic diary:local reactions; systemic events; use of antipyretic medication (up to 7 days after each vaccine dose).
Description: Safety population: participants who receive at least 1 dose of study vaccine. SAEs and AEs were grouped by system organ class and summarized. AEs included solicited AEs collected in electronic diary (local and systemic reactions; systematic assessment) and unsolicited events collected on case report form at each visit (nonsystematic assessment).
Groups:
- 13vPnC + DTaP - Infant Series: Participants who received 3 single 0.5 mL doses of 13vPnC subcutaneously 4 to 8 weeks apart along with 3 single 0.5 mL doses of DTaP subcutaneously (infant series), assessed from Infant Dose 1 through the blood draw 28 to 42 days post-infant series.
- 7vPnC + DTaP - Infant Series: Participants who received 3 single 0.5 mL doses of 7vPnC subcutaneously 4 to 8 weeks apart along with 3 single 0.5 mL doses of DTaP subcutaneously (infant series), assessed from Infant Dose 1 through the blood draw 28 to 42 days post-infant series.
- DTaP (Catch-up 7vPnC) - Infant Series: Participants who received 3 single 0.5 mL DTaP doses subcutaneously 4 to 8 weeks apart (infant series) followed by 2 single catch-up (CU) doses, CU Dose 1 and CU Dose 2 (separated by 4 to 6 weeks), of 7vPnC (Prevenar) 4 to 6 weeks post-infant series, assessed from Infant Dose 1 through the CU Dose 1.
- 13vPnC + DTaP - After the Infant Series; 7vPnC + DTaP - After the Infant Series: Participants who received 3 single 0.5 mL doses of 13vPnC subcutaneously 4 to 8 weeks apart along with 3 single 0.5 mL doses of DTaP subcutaneously (infant series), assessed after the infant series blood draw to the toddler dose.
- DTaP (Catch-up 7vPnC) - After the Infant Series: Participants who received 3 single 0.5 mL DTaP doses subcutaneously 4 to 8 weeks apart (infant series) followed by 2 single catch-up (CU) doses, CU Dose 1 and CU Dose 2 (separated by 4 to 6 weeks), of 7vPnC (Prevenar) 4 to 6 weeks post-infant series, assessed after CU Dose 1 to the toddler dose.
- 13vPnC + DTaP - Toddler Dose: Participants who received a single 0.5 mL dose of 13vPnC subcutaneously (toddler dose) along with 0.5 mL dose of DTaP subcutaneously, assessed from the toddler dose through the blood draw 28 to 42 days post-toddler dose.
- 7vPnC + DTaP - Toddler Dose: Participants who received a single 0.5 mL dose of 7vPnC subcutaneously (toddler dose) along with 0.5 mL dose of DTaP subcutaneously, assessed from the toddler dose through the blood draw 28 to 42 days post-toddler dose.
- DTaP (Catch-up 7vPnC) - Toddler Dose: Participants who received a single 0.5 mL DTaP dose subcutaneously (toddler dose) followed by a single catch-up (CU) dose (CU Dose 3) of 7vPnC (Prevenar) 4 to 6 weeks after toddler dose; assessed from toddler dose through the CU Dose 3.
- DTaP (Catch-up 7vPnC) - After the Toddler Dose: Participants who received a single 0.5 mL DTaP dose subcutaneously (toddler dose) followed by a single catch-up (CU) dose (CU Dose 3) of 7vPnC (Prevenar) 4 to 6 weeks after toddler dose; assessed after the CU Dose 3 to 28 to 42 days post-CU Dose 3.
Arm/Group | 13vPnC + DTaP - Infant Series | 7vPnC + DTaP - Infant Series | DTaP (Catch-up 7vPnC) - Infant Series | 13vPnC + DTaP - After the Infant Series | 7vPnC + DTaP - After the Infant Series | DTaP (Catch-up 7vPnC) - After the Infant Series | 13vPnC + DTaP - Toddler Dose | 7vPnC + DTaP - Toddler Dose | DTaP (Catch-up 7vPnC) - Toddler Dose | DTaP (Catch-up 7vPnC) - After the Toddler Dose
Serious Adverse Events (participants affected / at risk) | 5/183 | 8/183 | 10/183 | 13/183 | 15/183 | 10/183 | 0/162 | 4/162 | 2/169 | 2/169
Other Adverse Events (participants affected / at risk) | 147/183 | 160/183 | 155/183 | 20/183 | 27/183 | 147/183 | 104/162 | 99/162 | 112/169 | 105/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC + DTaP - Infant Series (N=183) | 7vPnC + DTaP - Infant Series (N=183) | DTaP (Catch-up 7vPnC) - Infant Series (N=183) | 13vPnC + DTaP - After the Infant Series (N=183) | 7vPnC + DTaP - After the Infant Series (N=183) | DTaP (Catch-up 7vPnC) - After the Infant Series (N=183) | 13vPnC + DTaP - Toddler Dose (N=162) | 7vPnC + DTaP - Toddler Dose (N=162) | DTaP (Catch-up 7vPnC) - Toddler Dose (N=169) | DTaP (Catch-up 7vPnC) - After the Toddler Dose (N=169)
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 1 | 1 | 6 | 5 | 3 | 0 | 3 | 1 | 2
Neuritis cranial (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Kawasaki's disease (Vascular disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Deafness bilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Exanthema subitum (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Herpangina (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mycoplasma infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rotavirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC + DTaP - Infant Series (N=183) | 7vPnC + DTaP - Infant Series (N=183) | DTaP (Catch-up 7vPnC) - Infant Series (N=183) | 13vPnC + DTaP - After the Infant Series (N=183) | 7vPnC + DTaP - After the Infant Series (N=183) | DTaP (Catch-up 7vPnC) - After the Infant Series (N=183) | 13vPnC + DTaP - Toddler Dose (N=162) | 7vPnC + DTaP - Toddler Dose (N=162) | DTaP (Catch-up 7vPnC) - Toddler Dose (N=169) | DTaP (Catch-up 7vPnC) - After the Toddler Dose (N=169)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 3 | 4 | 0 | 2 | 2 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blepharitis (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 7 | 11 | 20 | 0 | 0 | 9 | 2 | 3 | 2 | 6
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dacryostenosis acquired (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 7 | 5 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acetonaemic vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 4 | 3 | 3 | 0 | 5 | 0 | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 10 | 9 | 5 | 0 | 1 | 5 | 3 | 3 | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Application site erythema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site dermatitis (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 1 | 4 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 0
Injection site induration (General disorders) | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1
Pyrexia (General disorders) | 4 | 5 | 6 | 0 | 0 | 12 | 3 | 5 | 2 | 1
Vaccination site induration (General disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaccination site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaccination site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 2 | 2 | 2 | 6 | 3 | 6 | 2 | 0 | 1 | 0
Milk allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adenoviral conjunctivitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Adenovirus infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 2 | 2 | 5 | 0 | 0 | 2 | 0 | 1 | 1 | 1
Bronchitis (Infections and infestations) | 24 | 28 | 26 | 0 | 0 | 35 | 8 | 9 | 13 | 16
Candidiasis (Infections and infestations) | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 2
Conjunctivitis bacterial (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Conjunctivitis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 3 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Enteritis infectious (Infections and infestations) | 1 | 1 | 4 | 0 | 0 | 5 | 1 | 0 | 1 | 2
Echo virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema infectiosum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Exanthema subitum (Infections and infestations) | 10 | 17 | 19 | 0 | 0 | 22 | 6 | 3 | 3 | 4
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 28 | 24 | 31 | 0 | 0 | 30 | 3 | 7 | 5 | 9
Gastroenteritis norovirus (Infections and infestations) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 7 | 9 | 7 | 0 | 0 | 8 | 0 | 2 | 1 | 2
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Genital candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Genital infection fungal (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gianotti-Crosti syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 21 | 27 | 21 | 7
Herpangina (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 6 | 2
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Impetigo (Infections and infestations) | 3 | 3 | 2 | 0 | 0 | 4 | 1 | 4 | 4 | 2
Influenza (Infections and infestations) | 3 | 4 | 6 | 0 | 0 | 13 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Molluscum contagiosum (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 48 | 58 | 51 | 1 | 2 | 42 | 32 | 21 | 28 | 27
Omphalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 8 | 6 | 7 | 1 | 0 | 8 | 4 | 4 | 5 | 7
Otitis media acute (Infections and infestations) | 0 | 5 | 3 | 0 | 0 | 7 | 4 | 0 | 1 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 3 | 3 | 2 | 0 | 0 | 6 | 4 | 3 | 2 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus bronchitis (Infections and infestations) | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 9 | 14 | 4 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 2 | 3 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rotavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin candida (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 1 | 3 | 0 | 0 | 4 | 0 | 3 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 54 | 67 | 65 | 0 | 0 | 62 | 20 | 19 | 28 | 25
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 4 | 8 | 4 | 0 | 0 | 3 | 2 | 0 | 0 | 2
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Viral rash (Infections and infestations) | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 5 | 5
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 0
Chillblains (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Ear injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 1 | 2 | 1
Frostbite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Body height below normal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuritis cranial (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast swelling (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital labial adhesions (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Posthitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 10 | 5 | 6 | 15 | 1 | 2 | 0 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fibrinous bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infantile asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary artery stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 2 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Asteatosis (Skin and subcutaneous tissue disorders) | 8 | 7 | 5 | 1 | 3 | 2 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4 | 0 | 3 | 2 | 1 | 1 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 | 5 | 5 | 0 | 0 | 2 | 0 | 1 | 1 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 16 | 19 | 26 | 1 | 0 | 19 | 5 | 6 | 1 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 2 | 5 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 24 | 26 | 27 | 1 | 2 | 17 | 3 | 5 | 5 | 5
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 9 | 8 | 4 | 0 | 1 | 2 | 2 | 0 | 3 | 0
Eczema infantile (Skin and subcutaneous tissue disorders) | 12 | 7 | 7 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | 4 | 5 | 6 | 5 | 4
Hyperkeratosis palmaris and plantaris (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 2 | 5 | 0 | 0 | 2 | 2 | 3 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 5 | 4 | 0 | 0 | 4 | 2 | 2 | 1 | 2
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Kawasaki's disease (Vascular disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Redness (Any) (Skin and subcutaneous tissue disorders) | 100/171 | 96/172 | 17/165 | 0/0 | 0/0 | 0/0 | 92/148 | 87/152 | 52/149 | 0/0 — Infant Series Dose 1 and Toddler Dose
Redness (Any) (Skin and subcutaneous tissue disorders) | 104/166 | 104/168 | 59/161 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Redness (Any) (Skin and subcutaneous tissue disorders) | 90/168 | 83/162 | 36/156 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Redness (Mild) (Skin and subcutaneous tissue disorders) | 82/170 | 88/172 | 17/165 | 0/0 | 0/0 | 0/0 | 74/148 | 72/151 | 42/148 | 0/0 — Infant Series Dose 1 and Toddler Dose
Redness (Mild) (Skin and subcutaneous tissue disorders) | 93/166 | 95/167 | 56/161 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Redness (Mild) (Skin and subcutaneous tissue disorders) | 79/167 | 69/160 | 34/156 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 31/164 | 30/166 | 0/162 | 0/0 | 0/0 | 0/0 | 39/141 | 38/139 | 19/145 | 0/0 — Infant Series Dose 1 and Toddler Dose
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 41/157 | 43/159 | 13/156 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 26/152 | 34/154 | 3/153 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Redness (Severe) (Skin and subcutaneous tissue disorders) | 0/161 | 1/162 | 0/162 | 0/0 | 0/0 | 0/0 | 0/140 | 0/136 | 0/141 | 0/0 — Infant Series Dose 1 and Toddler Dose
Redness (Severe) (Skin and subcutaneous tissue disorders) | 0/157 | 0/154 | 0/154 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Redness (Severe) (Skin and subcutaneous tissue disorders) | 0/149 | 0/152 | 0/152 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Swelling (Any) (Skin and subcutaneous tissue disorders) | 69/168 | 60/168 | 8/164 | 0/0 | 0/0 | 0/0 | 73/149 | 66/144 | 39/148 | 0/0 — Infant Series Dose 1 and Toddler Dose
Swelling (Any) (Skin and subcutaneous tissue disorders) | 77/160 | 87/171 | 39/162 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Swelling (Any) (Skin and subcutaneous tissue disorders) | 72/164 | 59/157 | 34/159 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 64/168 | 53/168 | 8/164 | 0/0 | 0/0 | 0/0 | 63/147 | 60/143 | 33/146 | 0/0 — Infant Series Dose 1 and Toddler Dose
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 71/160 | 82/170 | 37/162 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 69/164 | 53/156 | 32/159 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 20/162 | 21/165 | 0/162 | 0/0 | 0/0 | 0/0 | 24/143 | 26/138 | 19/146 | 0/0 — Infant Series Dose 1 and Toddler Dose
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 31/157 | 28/157 | 9/155 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 16/150 | 23/154 | 4/153 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 0/161 | 1/162 | 0/162 | 0/0 | 0/0 | 0/0 | 0/140 | 0/136 | 0/141 | 0/0 — Infant Series Dose 1 and Toddler Dose
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 0/157 | 0/154 | 0/154 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 0/149 | 0/152 | 0/152 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 22/163 | 10/164 | 2/162 | 0/0 | 0/0 | 0/0 | 20/142 | 14/140 | 8/142 | 0/0 — Infant Series Dose 1 and Toddler Dose
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 23/159 | 7/154 | 3/155 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 12/153 | 11/155 | 4/153 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 0/161 | 0/162 | 0/162 | 0/0 | 0/0 | 0/0 | 1/140 | 0/136 | 0/141 | 0/0 — Infant Series Dose 1 and Toddler Dose
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 1/157 | 0/154 | 0/154 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 0/149 | 0/152 | 1/152 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Fever >=37.5, =<39 degrees C (General disorders) | 61/168 | 57/168 | 36/165 | 0/0 | 0/0 | 0/0 | 71/145 | 72/146 | 46/146 | 0/0 — Infant Series Dose 1 and Toddler Dose
Fever >=37.5, =<39 degrees C (General disorders) | 61/166 | 59/161 | 34/155 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Fever >=37.5, =<39 degrees C (General disorders) | 56/162 | 49/161 | 38/157 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Fever >=39, =<40 degrees C (General disorders) | 1/161 | 2/163 | 1/162 | 0/0 | 0/0 | 0/0 | 6/141 | 12/136 | 5/141 | 0/0 — Infant Series Dose 1 and Toddler Dose
Fever >=39, =<40 degrees C (General disorders) | 3/158 | 6/155 | 1/154 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Fever >=39, =<40 degrees C (General disorders) | 5/150 | 3/152 | 5/153 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Fever >40 degrees C (General disorders) | 0/161 | 0/162 | 0/162 | 0/0 | 0/0 | 0/0 | 2/139 | 3/137 | 0/141 | 0/0 — Infant Series Dose 1 and Toddler Dose
Fever >40 degrees C (General disorders) | 0/157 | 0/154 | 0/154 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Fever >40 degrees C (General disorders) | 0/149 | 1/152 | 0/152 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Decreased appetite (General disorders) | 21/163 | 15/163 | 12/165 | 0/0 | 0/0 | 0/0 | 28/143 | 28/141 | 14/143 | 0/0 — Infant Series Dose 1 and Toddler Dose
Decreased appetite (General disorders) | 18/158 | 23/159 | 11/155 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Decreased appetite (General disorders) | 15/152 | 15/155 | 9/154 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Irritability (General disorders) | 31/165 | 27/164 | 20/164 | 0/0 | 0/0 | 0/0 | 26/143 | 30/141 | 24/144 | 0/0 — Infant Series Dose 1 and Toddler Dose
Irritability (General disorders) | 29/162 | 29/155 | 17/156 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Irritability (General disorders) | 27/154 | 23/156 | 18/154 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Increased sleep (General disorders) | 49/170 | 44/165 | 36/165 | 0/0 | 0/0 | 0/0 | 27/145 | 25/142 | 23/143 | 0/0 — Infant Series Dose 1 and Toddler Dose
Increased sleep (General disorders) | 37/163 | 35/158 | 37/163 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Increased sleep (General disorders) | 31/151 | 32/157 | 23/154 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Decreased sleep (General disorders) | 30/164 | 36/169 | 23/167 | 0/0 | 0/0 | 0/0 | 18/142 | 13/137 | 16/141 | 0/0 — Infant Series Dose 1 and Toddler Dose
Decreased sleep (General disorders) | 30/161 | 19/157 | 19/157 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Decreased sleep (General disorders) | 28/154 | 20/156 | 15/153 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Hives (urticaria) (General disorders) | 5/161 | 2/162 | 0/162 | 0/0 | 0/0 | 0/0 | 5/140 | 3/136 | 3/141 | 0/0 — Infant Series Dose 1 and Toddler Dose
Hives (urticaria) (General disorders) | 4/157 | 2/154 | 3/154 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Hives (urticaria) (General disorders) | 2/149 | 0/152 | 2/152 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Use of antipyretic medication to treat symptoms (General disorders) | 6/161 | 4/162 | 1/162 | 0/0 | 0/0 | 0/0 | 10/141 | 13/138 | 6/142 | 0/0 — Infant Series Dose 1 and Toddler Dose
Use of antipyretic medication to treat symptoms (General disorders) | 5/160 | 7/155 | 2/154 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Use of antipyretic medication to treat symptoms (General disorders) | 3/150 | 5/153 | 7/154 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.